CLINICAL TRIAL: NCT01856244
Title: Sensorimotor Treadmill Training to Improve Gait and Balance in Parkinson's Disease
Brief Title: Stability and Balance in Locomotion Through Exercise
Acronym: StaBLE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: German Foundation for Neurology (Other); Department of Molecular Neurology, Faculty of Medicine, University Erlangen-Nürnberg (Other)
Responsible Party: Principal Investigator, Prof. Dr. Klaus Pfeifer, Prof. Dr., University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DSN-0613
Record Dates: First submitted 2013-05-08; First posted 2013-05-17 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; treadmill training; gait; balance; mobility
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sensorimotor treadmill training (Experimental): specific treadmill control using oscillating platform
  Interventions: Behavioral: treadmill walking; Device: Treadmill
- conventional treadmill training (Active Comparator): conventional treadmill control
  Interventions: Behavioral: treadmill walking; Device: Treadmill

INTERVENTIONS:
Behavioral: treadmill walking
Device: Treadmill

SUMMARY:
Persons with Morbus Parkinson commonly develop gait and balance disorders leading to dependence, loss of mobility and a high risk of falling.

This study investigates the effectiveness of a sensorimotor treadmill intervention to improve walking and balance abilities in persons with early stages of Parkinson's disease. The sensorimotor treadmill training is conducted on a special treadmill device which is challenging the participants by small oscillations. This intervention, which is supposed to simulate walking on natural, uneven surfaces, is compared to a conventional treadmill training.

Hypothesis: Sensorimotor treadmill training leads to larger improvements in walking and balance abilities as compared to conventional treadmill exercise.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease stage 1-3 Hoehn and Yahr
* United Parkinson Disease Rating Scale (UPDRS) 'gait' or 'postural stability' subscore of 1 or more
* Ability to stand unaided and walk without an assistive device
* Stable medication during the study period

Exclusion Criteria:

* On-off and wearing-off phenomena
* Unstable medical or psychiatric illness
* Clinically relevant cardiovascular or orthopaedic disease
* Severe polyneuropathy
* Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Gait Speed | 8 weeks and 20 weeks
  Self selected walking speed is assessed on a 10 meter walk distance
Change from Baseline Balance | 8 weeks and 20 weeks
  Mini - Balance Evaluation Systems Test (Mini - BESTest), Postural Sway in the Romberg Test with eyes open and eyes closed for 30 seconds

SECONDARY OUTCOMES:
Change from Baseline Gait Performance | 8 weeks and 20 weeks
  Two Minute Walk Test (2MWT), Timed "up-and-go" Test, Assessment of tempo-spatial gait parameters
Change from Baseline Mobility | 8 weeks and 20 weeks
  Rivermead Mobility Index
Change from Baseline Unified Parkinson's Disease Rating Scale (UPDRS) | 8 weeks and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Pfeifer, Prof. Dr., Principal Investigator — Friedrich-Alexander-Universität Erlangen-Nürnberg (FAU), Institute of Sport Science and Sport
Locations (1):
- Friedrich-Alexander-Universität Erlangen-Nürnberg (FAU), Institute of Sport Science and Sport, Gebbertstr. 123b, Erlangen, Germany

REFERENCES:
- [Background] Klamroth S, Steib S, Devan S, Pfeifer K. Effects of Exercise Therapy on Postural Instability in Parkinson Disease: A Meta-analysis. J Neurol Phys Ther. 2016 Jan;40(1):3-14. doi: 10.1097/NPT.0000000000000117. PMID 26655098
- [Result] Klamroth S, Steib S, Gassner H, Gossler J, Winkler J, Eskofier B, Klucken J, Pfeifer K. Immediate effects of perturbation treadmill training on gait and postural control in patients with Parkinson's disease. Gait Posture. 2016 Oct;50:102-108. doi: 10.1016/j.gaitpost.2016.08.020. Epub 2016 Aug 26. PMID 27591395